CLINICAL TRIAL: NCT06177886
Title: Incidence and Predictive Risk Factors of Acute Kidney Injury in Pediatric Polytrauma Patients Admitted to Assiut University Trauma Unit: a Cross-sectional Study
Brief Title: Acute Kidney Injury in Pediatric Polytrauma Patients at Assiut University Trauma Unit: A Cross-Sectional Study on Incidence and Predictive Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Atef Alsayed, resident doctor at emergency medicine department, Assiut University
Other Study IDs: AKIPPP
Record Dates: First submitted 2023-12-02; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the true incidence and clinical presentation of post-traumatic AKI in hospitalized pediatric patients and identify the risk, and severity of AKI. The results would aid the emergency physicians in the early identification of those at risk of AKI to establish a resuscitation strategy that aims at preventing AKI

DETAILED DESCRIPTION:
Trauma is a leading cause of morbidity and mortality throughout Africa and the leading cause of mortality worldwide for children and young adults (5-29 years of age).

Organ failure, including AKI, is the third leading cause of mortality in trauma patients, after bleeding and brain injuries.

Trauma patients are at risk of AKI caused by renal hypoperfusion (secondary to haemorrhagic shock), rhabdomyolysis, direct renal injury, abdominal compartment syndrome, or the nephrotoxic effects of therapies.

The majority of trauma-based AKI studies worldwide have looked at critically ill adult trauma patients and these report highly variable AKI rates, ranging 1-50%.

Though pediatric trauma studies on AKI are scarce, a California study suggests 13% of pediatric post-traumatic rhabdomyolysis patients experience AKI.

Acute kidney injury (AKI) is described as a spectrum of abruptly compromised renal functions that result in impaired balance of fluid, electrolytes, and waste products. It is recognized as an increasingly common cause of morbidity and mortality in children.

AKI is defined according to The Kidney Disease: Improving Global Outcomes (KDIGO) Clinical Practice Guidelines as any of the following: increase in serum creatinine by ≥0.3 mg/dL within 48 h; or increase in serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior seven days; or urine volume <0.5ml /kg/ h for 6 hr.

Preventive measures for AKI are currently the mainstay of non-dialytic AKI management. They include the use of a pediatric early warning score for early detection of AKI, preparation to provide for volume resuscitation in patients with hypovolemia related oliguria, and halting the administration of angiotensin converting enzyme inhibitors and angiotensin II receptor blockers in such patients until their volume status is stabilized. Using appropriate nephrotoxic drug doses (i.e., vancomycin and/or contrast media) to reduce harm to the kidneys.

RRT is the most effective way of managing severe AKI. Peritoneal dialysis has shown as an effective adjuvant treatment for achieving a negative fluid balance, decreasing mechanical ventilation duration, and reducing electrolyte disturbances There is currently no specific effective treatment after the occurrence of established AKI Early detection and prevention of AKI is essential.

ELIGIBILITY:
Inclusion Criteria:

* The present study will be conducted on pediatric patients with multiple traumas of both genders aged 2yr to 18 yr who have no previous history of kidney disease or chronic illness.

Exclusion Criteria:

* Patients who are less than 2 years old or more than 18 years old.
* Direct trauma kidney or localized individual trauma
* children with preexisting kidney disease
* children with drug nephrotoxicity
* children underwent renal transplant
* children post-cardiac arrest
* Patients leaving the hospital on the same day or transferred to a different hospital will be excluded from this study.
* Patients refusing the study will be excluded.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From September 2023 till September 2024, all patients admitted to the emergency department who meet the eligibility criteria will be recruited in this study after obtaining informed consent from their legal guardians.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AKI in Pediatric Trauma Patients Admitted to ER | baseline
  Describing the true incidence of AKI in pediatric trauma patients who are admitted to ER.
  a) Identification of AKI according to the KDIGO guidelines as follows: I. Increase in serum creatinine by ≥0.3 mg/dL (≥26.5 micromol/L) within 48 hours, or II. Increase in serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior seven days, or III. Urine volume <0.5 mL/kg/hour for six hours
timing of AKI in pediatric trauma patients admitted to ER | baseline
  time period between admission and diagnosis of AKI

SECONDARY OUTCOMES:
Risk Identification of AKI in pediatric trauma patients | baseline
  Identifying risk for AKI as presence of shock and/or rhabdomyolysis. Exposure to nephrotoxic drugs .
mortality outcomes of AKI in pediatric trauma patients | Baseline
  The standardized mortality ratio represents the excess mortality and will be calculated using the observed number of lethal cases divided by the predicted number of lethal cases. The observed count will be obtained from the study data. The predicted number will be obtained by implementing the percentage of mortality risk from all the tools used. The individual values of the risk scores will be averaged to represent the study population.

REFERENCES:
- [Background] Harrois A, Soyer B, Gauss T, Hamada S, Raux M, Duranteau J; Traumabase(R) Group. Prevalence and risk factors for acute kidney injury among trauma patients: a multicenter cohort study. Crit Care. 2018 Dec 18;22(1):344. doi: 10.1186/s13054-018-2265-9. PMID 30563549
- [Background] Harrois A, Libert N, Duranteau J. Acute kidney injury in trauma patients. Curr Opin Crit Care. 2017 Dec;23(6):447-456. doi: 10.1097/MCC.0000000000000463. PMID 29035925
- [Background] Reilly JP, Anderson BJ, Mangalmurti NS, Nguyen TD, Holena DN, Wu Q, Nguyen ET, Reilly MP, Lanken PN, Christie JD, Meyer NJ, Shashaty MG. The ABO Histo-Blood Group and AKI in Critically Ill Patients with Trauma or Sepsis. Clin J Am Soc Nephrol. 2015 Nov 6;10(11):1911-20. doi: 10.2215/CJN.12201214. Epub 2015 Sep 4. PMID 26342043
- [Background] Bagshaw SM, George C, Gibney RT, Bellomo R. A multi-center evaluation of early acute kidney injury in critically ill trauma patients. Ren Fail. 2008;30(6):581-9. doi: 10.1080/08860220802134649. PMID 18661407
- [Background] Eriksson M, Brattstrom O, Martensson J, Larsson E, Oldner A. Acute kidney injury following severe trauma: Risk factors and long-term outcome. J Trauma Acute Care Surg. 2015 Sep;79(3):407-12. doi: 10.1097/TA.0000000000000727. PMID 26307873
- [Background] Fujinaga J, Kuriyama A, Shimada N. Incidence and risk factors of acute kidney injury in the Japanese trauma population: A prospective cohort study. Injury. 2017 Oct;48(10):2145-2149. doi: 10.1016/j.injury.2017.08.022. Epub 2017 Aug 15. PMID 28842286
- [Background] Santos PR, Monteiro DL. Acute kidney injury in an intensive care unit of a general hospital with emergency room specializing in trauma: an observational prospective study. BMC Nephrol. 2015 Mar 19;16:30. doi: 10.1186/s12882-015-0026-4. PMID 25885883
- [Background] Talving P, Karamanos E, Skiada D, Lam L, Teixeira PG, Inaba K, Johnson J, Demetriades D. Relationship of creatine kinase elevation and acute kidney injury in pediatric trauma patients. J Trauma Acute Care Surg. 2013 Mar;74(3):912-6. doi: 10.1097/TA.0b013e318278954e. PMID 23425757
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] National Clinical Guideline Centre (UK). Acute Kidney Injury: Prevention, Detection and Management Up to the Point of Renal Replacement Therapy [Internet]. London: Royal College of Physicians (UK); 2013 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK247665/ PMID 25340231
- [Background] Ricci Z, Romagnoli S. Prescription of dialysis in pediatric acute kidney injury. Minerva Pediatr. 2015 Apr;67(2):159-67. Epub 2015 Jan 23. PMID 25615028
- [Background] Kwiatkowski DM, Goldstein SL, Cooper DS, Nelson DP, Morales DL, Krawczeski CD. Peritoneal Dialysis vs Furosemide for Prevention of Fluid Overload in Infants After Cardiac Surgery: A Randomized Clinical Trial. JAMA Pediatr. 2017 Apr 1;171(4):357-364. doi: 10.1001/jamapediatrics.2016.4538. PMID 28241247
- [Background] Kwiatkowski DM, Menon S, Krawczeski CD, Goldstein SL, Morales DL, Phillips A, Manning PB, Eghtesady P, Wang Y, Nelson DP, Cooper DS. Improved outcomes with peritoneal dialysis catheter placement after cardiopulmonary bypass in infants. J Thorac Cardiovasc Surg. 2015 Jan;149(1):230-6. doi: 10.1016/j.jtcvs.2013.11.040. Epub 2013 Dec 31. PMID 24503323
- [Background] Bojan M, Gioanni S, Vouhe PR, Journois D, Pouard P. Early initiation of peritoneal dialysis in neonates and infants with acute kidney injury following cardiac surgery is associated with a significant decrease in mortality. Kidney Int. 2012 Aug;82(4):474-81. doi: 10.1038/ki.2012.172. PMID 22622499
- [Background] Webb TN, Goldstein SL. Congenital heart surgery and acute kidney injury. Curr Opin Anaesthesiol. 2017 Feb;30(1):105-112. doi: 10.1097/ACO.0000000000000406. PMID 27748669
- [Background] Kellum JA, Bellomo R, Ronco C. Classification of acute kidney injury using RIFLE: What's the purpose? Crit Care Med. 2007 Aug;35(8):1983-4. doi: 10.1097/01.CCM.0000277518.67114.F8. No abstract available. PMID 17667247
- [Background] de Abreu KL, Silva Junior GB, Barreto AG, Melo FM, Oliveira BB, Mota RM, Rocha NA, Silva SL, Araujo SM, Daher EF. Acute kidney injury after trauma: Prevalence, clinical characteristics and RIFLE classification. Indian J Crit Care Med. 2010 Jul;14(3):121-8. doi: 10.4103/0972-5229.74170. PMID 21253345
- [Background] Li J, Han B, Li H, Deng H, Mendez-Sanchez N, Guo X, Qi X. Association of coagulopathy with the risk of bleeding after invasive procedures in liver cirrhosis. Saudi J Gastroenterol. 2018 Jul-Aug;24(4):220-227. doi: 10.4103/sjg.SJG_486_17. PMID 29956689